CLINICAL TRIAL: NCT03565172
Title: Efficacy of a Long Term, High Intensity and Long Time Stretch Training Program on Viscoelasticity Plantarflexors Muscle in Children With Cerebral Palsy (CP).
Acronym: LONGSTRETCH PC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: protocol with too many constraints. long protocol
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18CH033; ID-RCB (Other: 2018-A00709-46)
Record Dates: First submitted 2018-06-12; First posted 2018-06-21 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Palsy, Spastic; Children, Only
Keywords: cerebral palsy; stretching; isokinetic dynamometer; ultrasound; ankle; children
MeSH Terms: conditions — Cerebral Palsy | interventions — Ultrasonography; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: The methodology used is : Single Case Experimental Design (SCED).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with spastic cerebral palsy (Experimental): Children with spastic cerebral palsy will be included. They will have 3 phases:
  * Baseline: 4, 5 or 6 evaluations
  * Intervention: 9 evaluations before and after every stretching session
  * Follow-up: 4, 5 or 6 evaluations
  The evaluation part will be composed of isokinetic dynamometer with ultrasound and Visual Analog Scale (VAS). The number of evaluations at baseline and follow-up will be randomized before the study by Single Case Experimental Design (SCED) methodology.
  Interventions: Diagnostic Test: isokinetic dynamometer with ultrasound; Other: Visual Analog Scale (VAS); Diagnostic Test: Stretching

INTERVENTIONS:
Diagnostic Test: isokinetic dynamometer with ultrasound — children are lying prone on a isokinetic dynamometer with ultrasound which stretches spastic and paretic plantarflexors muscles very slowly until maximal torque tolerated. The parameters can be measured.
Other: Visual Analog Scale (VAS) — the discomfort level will be measured by Visual Analog Scale (VAS) completed by children. 0 = no discomfort and 10 = maximum discomfort
Diagnostic Test: Stretching — the ankle of children will be mobilized for 5 minutes (first two weeks) to 10 minutes (last two weeks).

SUMMARY:
Children with cerebral palsy present early in the childhood altered muscular properties, as soon as structural or stiffness. In the gastrocnemius muscle, altered muscular properties are characterized by short muscle belly length and increased stiffness which contribute to contracture and limiting joint range of motion.

DETAILED DESCRIPTION:
This study assess efficacy of a long term stretching program of plantarflexors muscle on their viscoelasticity properties and maximal dorsiflexion angle gain. Stretching program is characterized by 3 phases: baseline, intervention and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 16 years
* Children diagnosed spastic cerebral palsy
* Children with decrease maximal dorsiflexion angle under +5° in the last four weeks
* Children who don't understand instructions

Exclusion Criteria:

* Children who had damage orthopedics or surgical operation contraindicating realization of the experimental protocol
* Hospitalization incompatible with the progress of the protocol.
* Children who had botulinum injection, extensions casts or the implementation of new equipment (night or day orthosis) for less than three months or the progress of the protocol.
* Children having analgesic treatment in progress

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
slope of the torque-angle curve | up to 12 weeks
  Analysis of the slope of the torque-angle curve in Nm/°. It is measured by isokinetic dynamometer with ultrasound.

SECONDARY OUTCOMES:
Maximal dorsiflexion angle | up to 12 weeks
  Analysis of the maximal dorsiflexion angle in degrees. It is measured by isokinetic dynamometer with ultrasound.
Slope of the torque- MyoTendinous Junction (MTJ) displacement | up to 12 weeks
  Analysis of the Slope of the torque- MyoTendinous Junction (MTJ) displacement in cm/°.
  It is measured by isokinetic dynamometer with ultrasound.
MyoTendinous Junction (MTJ) displacement of muscle triceps sural | up to 12 weeks
  Analysis of the MyoTendinous Junction (MTJ) displacement of muscle triceps sural in cm.
  It is measured by isokinetic dynamometer with ultrasound.
muscle triceps sural, muscle body of the medial gastrocnemius muscle and Achilles tendon | up to 12 weeks
  Correlation of the length of Musculo-Tendinous Unit (MTU) of muscle triceps sural, muscle body of the medial gastrocnemius muscle and Achilles tendon.
  It is measured by isokinetic dynamometer with ultrasound.
discomfort level | up to 12 weeks
  Analysis of the discomfort level. It is measured by Visual Analog Scale (VAS) completed by children. 0 = no discomfort and 10 = maximum discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GAUTHERON, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No